CLINICAL TRIAL: NCT05710159
Title: The iBlad App - a National, Exploratory Study on a Multimodality Smartphone App in Bladder Cancer for Better Understanding of Symptoms, Quality of Life and Need for Supportive Care
Brief Title: The iBlad App - a National, Exploratory Study on a Multimodality Smartphone App for Bladder Cancer Patients
Acronym: iBLAD-app
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Laerke Kjaer Tolstrup, RN, PhD, Odense University Hospital
Other Study IDs: R261-A16126
Record Dates: First submitted 2022-12-07; First posted 2023-02-02 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: iBLAD Application to monitor symptoms and quality of life by the use of pateint-reported outcomes — Development and implementation of a national multimodality application for patients with bladder cancer that builds upon knowledge from the iBLAD study.

SUMMARY:
The aims of this project are:

* to develop and implement a national multimodality application for patients with bladder cancer that builds upon knowledge from the iBLAD study.
* to investigate how the app, containing PRO questions on symptoms and QoL, information for health care providers, and peer-to-peer advice, can provide more knowledge on symptoms, QoL, and the need for supportive care.
* to examine the usability of and patient satisfaction with the app using qualitative methods.

DETAILED DESCRIPTION:
Design The iBLAD app study is an investigator-initiated, national, Danish multicenter, exploratory trial connected to the group of bladder cancer responsible specialists at the six Danish treatment centers. The study is carried out in accordance with the SPIRIT-PRO Protocol Guidance.

Study plan The app is developed by the app provider Journl who is specialized in ePRO apps. The app is in Danish. The patient will be able to download the app and create a user profile when a clinician has registered the patient in Journl's system as a bladder cancer patient in oncological treatment. After giving informed consent, the patient will (be helped to) download the app on their private smartphone. The patient will answer the first questionnaires in relation to the first treatment. The first patient is expected to be enrolled in December 2022. Patients can use the app as long as treatment is ongoing. Patients can at any time withdraw their consent and stop using the app. The patient will receive daily notifications from the app if there is an unanswered questionnaire to minimize missing data.

Questionnaires In the app, Bladder cancer patients will receive an electronic questionnaire weekly with selected questions from the PRO-CTCAE library. The questions have been carefully selected for their specific disease and condition. The epo-CTCAE questionnaire consists of 15 symptoms comprising of 30 questions on symptoms and side effects. Each symptom is elicited using between one to three questions on frequency, severity, and interference with daily activities. Weekly reporting was chosen as this is the preferred recall period for PRO-CTCAE questionnaires. Depending on the patients´ response and due to predefined thresholds, the patient will get feedback for supportive care or be advised to contact the hospital. Moreover, the patients will be asked to complete EORTC QLQ-C30 and EORTC QLQ-BLM30 monthly to monitor their QoL (see supplementary material). All electronic questionnaires will be completed at home. An expert group, consisting of nurses and clinicians, has selected the questionnaires as the most relevant questionnaires for this patient population.

Patient feedback and inclusion in the clinical encounter The questionnaires are the same regardless of the patient's oncological treatment but is developed to cover both chemotherapy and ICI. The patients receive immediate feedback in the app as they complete the symptom questionnaire. The advice given can continuously be found in the app. The advice is based on an algorithm linked to the severity of the symptoms or side effects that the patient reports. The algorithm including type of intervention was developed by the expert group. The symptom and QoL scores are also sent to the hospital where the clinician can access the patient reporting and are trained and prompted to review the scores at patient visits. Thus, the patient reporting not only serves as a reflection of the patient's condition to be used for research purposes but can also be used as a dialogue tool during the clinical encounter. Accordingly, the app will enable regular symptom tracking, feedback to patients and QoL reporting to achieve earlier symptom management and improved supportive care. The ePRO questionnaires are added to standard of care and the symptoms highlighted will be treated in alignment with standard procedures. In routine care, clinicians carry out toxicity registration prior to each cycle of anti-neoplastic treatment, typically every three or four weeks. The weekly patient reporting in the app takes place at home in between visits to the hospital. Alert algorithms and thresholds for alerts can be seen in Supplementary material.

Patient videos In addition to completing questionnaires in the app, the patients will also gain access to a variety of short videos with former bladder patients recruited from the Danish bladder cancer organization. The subjects of the videos were decided on during a workshop carried out with six bladder cancer patients who had all received anti-neoplastic treatment. Thus, the participants in the workshop took part in deciding what the app should contain in terms of informative and relevant video material on the experiences of bladder cancer patients. Fifty-three videos will be produced with five bladder cancer patients (three men and two women). In the videos, the patients share peer-to-peer insights on how they experience being bladder cancer patients, covering a wide range of topics such as living with cancer, operation, treatment, sexual issues, family relations, rehabilitation and quality of life.

Evaluation Patients will receive questionnaires on symptoms and QoL as long as treatment is ongoing. After 4 weeks of treatment, the patients will be asked to complete a validated Patient-Reported Experience Measure in the clinic to evaluate acceptability of the app. In addition, individual interviews will be performed with participants in the study from all six centers where usability and patient satisfaction is evaluated.

Endpoints Primary outcome is PRO symptoms´ correlation to QoL measured by EORTC-QLQ-C30 and the specific bladder cancer questionnaire EORTC-QLQ-BLM-30 and submodules of these. Additionally, specific PRO symptoms development over time and time-dependency in relation to QoL will be investigated. The study is non-comparative and analyses will be exploratory. Secondary endpoints will be level of user acceptability and patient satisfaction.

Sample size No sample size calculation has been performed due to the study's explorative nature. To secure a broad geographic representation the aim is to include at least 100 patients with a minimum of 10 patients from each of the six centers. The study will be analyzed when 100 patients have been followed for at least 3 months. An interim analyses will be performed after 30 included patients primarily to evaluate compliance and adherence to the app.

Data collection and statistics Information on age, time of diagnosis, gender, histology, TNM stage, treatment type, treatment line and performance status will be noted. A baseline questionnaire on symptoms and QoL will be completed. The analyses of ePRO data will include descriptive statistics for both changes from baseline and observed scores after 1, 2, 3, 4, 5 and 6 months of participation in the study. In case of missing data, imputation will not take place. PRO-data will be monitored regularly, in the beginning on a weekly basis. After 12 weeks, we will shift to monthly monitoring if adherence is acceptable. If patients do not comply with the study protocol, they will be contacted by the project manager and/or withdrawn from the study. Eligible patients will be informed about this upon enrolment and that it will have no impact on their treatment.

Ethics declaration The iBLAD app study was exempt for review by the Medical Research Ethics Committee, will follow General Data Protection Regulation, and is registered at the Capital Region of Denmark. The results of the study will be reported in a scientific journal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bladder cancer defined as both urothelial tract-, bladder- and urethral cancer initiating first or second-line standard therapy with either chemotherapy or immunotherapy
* Age ≥ 18 years,
* Performance status ≤ 2
* Ability to read Danish
* No serious cognitive impairment
* Informed consent.

Exclusion Criteria:

* No smartphone,
* Dementia, mental alteration, or psychiatric disease that can compromise informed consent from the patient and/or adherence to the protocol and the monitoring of the trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bladder cancer defined as both urothelial tract-, bladder- and urethral cancer initiating first or second-line standard therapy with either chemotherapy or immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Development and implementation of the iBLAD-app | 2 years
  To develop and implement a national multimodality application (app) for patients with bladder cancer t

SECONDARY OUTCOMES:
App contributions | 2 years
  To investigate how the app, containing PRO questions on symptoms and QoL, information for health care providers, and peer-to-peer advice, can provide more knowledge on symptoms, QoL, and the need for supportive care.
Usability and evaluation | 2 years
  To examine the usability of and patient satisfaction with the app using qualitative methods.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Pappot, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Taarnhoj GA, Lindberg H, Johansen C, Pappot H. Patient-Reported Outcomes, Health-Related Quality of Life, and Clinical Outcomes for Urothelial Cancer Patients Receiving Chemo- or Immunotherapy: A Real-Life Experience. J Clin Med. 2021 Apr 24;10(9):1852. doi: 10.3390/jcm10091852. PMID 33923176
- [Background] Taarnhoj GA, Johansen C, Lindberg H, Basch E, Dueck A, Pappot H. Patient reported symptoms associated with quality of life during chemo- or immunotherapy for bladder cancer patients with advanced disease. Cancer Med. 2020 May;9(9):3078-3087. doi: 10.1002/cam4.2958. Epub 2020 Mar 10. PMID 32154663
- [Background] Taarnhoj GA, Lindberg H, Dohn LH, Omland LH, Hjollund NH, Johansen C, Pappot H. Electronic reporting of patient-reported outcomes in a fragile and comorbid population during cancer therapy - a feasibility study. Health Qual Life Outcomes. 2020 Jul 11;18(1):225. doi: 10.1186/s12955-020-01480-3. PMID 32653005
- [Background] Taarnhoj GA, Lindberg H, Johansen C, Pappot H. Patient-reported outcomes item selection for bladder cancer patients in chemo- or immunotherapy. J Patient Rep Outcomes. 2019 Aug 22;3(1):56. doi: 10.1186/s41687-019-0141-2. PMID 31440865